CLINICAL TRIAL: NCT03440333
Title: A Multicenter Study of Pulmonary Surfactant(PS) Therapy in the Treatment of Neonatal Acute Respiratory Distress Syndrome(RDS) at High Altitude Area
Brief Title: Pulmonary Surfactant(PS) Therapy at High Altitude Area
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: the first people hospital of Tibet autonomous region (Unknown); the second people hospital of Lasa (Unknown); the first people hospital of Shigatse (Unknown); the first people hospital of Lasa (Unknown); the people hospital of Linzhi (Unknown); the people hospital of Laqu (Unknown); Shannan People's Hospital (Other); the people hospital of Changdu (Unknown); the people hospital of Ali (Unknown); the second people hospital of Tibet autonomous region (Unknown); Women and Children Hospital of Qinghai Province (Other)
Responsible Party: Principal Investigator, Ma Juan, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: pulmonary surfactant(PS)
Record Dates: First submitted 2018-02-03; First posted 2018-02-22 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: NRDS; Surfactant
MeSH Terms: interventions — Surface-Active Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: surfactant — Pulmonary surfactant was administrated if the baby was diagnosed with respiratory distress syndrome

SUMMARY:
The traditional concept believes that the etiology of neonatal respiratory distress syndrome (RDS) is immature development of lung,especially the surfactant synthesis system,and RDS is still one of the major causes of mortality and morbidity in newborns, especially premature infants[1].In recent years, using pulmonary surfactant replacement therapy (PS treatment) in the treatment of respiratory distress syndrome (RDS) is a major breakthrough in neonatal medicine [2].Combined with clinical practice and experience,and through Meta analysis of related randomized controlled trials (RCTs),it confirms that natural surfactant treatment can reduce mortality,the incidence of pulmonary air leaks (pneumothorax and interstitial lung emphysema),and the incidence of bronchopulmonary dysplasia (BPD) or 28-day-old mortality.For RDS in preterm infants whose gestation is <35 weeks ,surfactant replacement therapy is also more effective than in nearly term and full term infants.Therefore, in the analysis of cases of different gestational age groups,the investigators should focus on the study of premature infants cases.Due to less relevant research for using PS treatment to cure newborn RDS in high altitude area,this retrospective study conducts statistics and analysis of recently three-year cases in some hospital of high altitude area,to explore the treatment effect of the high altitude region and the impact of altitude on the treatment.

DETAILED DESCRIPTION:
in order to explore feasibility and efficacy for PS treatment of newborn RDS in high-altitude area ,and its efficacy at different altitudes, the investigators conduct a multi-center retrospective study of RDS cases in Qinghai and Tibet these two high-altitude area,and use RDS cases under the unique conditions to do statistics and analysis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with respiratory distress syndrome(RDS)

Exclusion Criteria:

* major congenital abnormalities

Ages: 1 Minute to 12 Hours | Sex: All
Age Groups: Child
Study Population: the preterm infants less than 37 weeks were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
the intubation rate | one week
  the effect of PS treatment for NRDS
the incidence of NRDS in different altitudes | one week
  different altitudes may result in different rate of NRDS